CLINICAL TRIAL: NCT01864850
Title: Non Inferiority Randomized Trial of Standard Radiotherapy Versus Hypofractionated Split Course Radiotherapy in Elderly Vulnerable Patients With Inoperable Head and Neck Squamous Cell Carcinoma
Brief Title: Non Inferiority Trial of Standard RT Versus Hypofractionated Split Course in Elderly Vulnerable Patients With HNSCC
Acronym: ELAN-RT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GORTEC ELAN-RT
Record Dates: First submitted 2013-05-21; First posted 2013-05-30 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Elderly; Geriatry
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Radiotherapy
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard RT (Active Comparator): 70 Gy / 7 weeks / 2 Gy per fraction
  Interventions: Radiation: Standard RT
- Hypofractionated RT (Experimental): 55 Gy / 7 weeks with 2 weeks interruption / 3 Gy per fraction until 30 Gy, after interruption 2.5 Gy per fraction until 55 Gy
  Interventions: Radiation: Hypofractionated RT

INTERVENTIONS:
Radiation: Standard RT — 70 Gy / 7 weeks / 2 Gy per fraction
  Arms: Standard RT
Radiation: Hypofractionated RT — 55 Gy / 7 weeks with 2 weeks interruption / 3 Gy per fraction until 30 Gy, after interruption 2.5 Gy per fraction until 55 Gy
  Arms: Hypofractionated RT

SUMMARY:
Randomized comparison between standard radiotherapy and hypofractionated split course schedule. Compared to standard radiotherapy, the investigators expect that hypofractionated split course (interruption of 2 weeks) radiotherapy will improve compliance to treatment, acute tolerance of treatment, preservation of autonomy, prevention of malnutrition, with the same efficacy, measured by the locoregional control rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 or over
* SIOG group 2 (vulnerable)
* Life expectancy > 12 weeks
* PS < 2
* Histologically confirmed diagnosis of squamous cell carcinoma of head and neck: oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, cervical nodes (unknown primary).
* First line treatment
* At least one measurable lesion (RECIST)
* Stage II to IV
* Patients unsuitable for surgery of the primary tumour: non resectable tumor, anesthesia contra indication, patient's refusal, or organ sparing approach. Cervical nodes dissection authorized
* Patients planned to be treated in a curative intent with radiotherapy alone on primary tumor site and on at least one head and neck node area
* Consent form signed

Exclusion Criteria:

* Primary squamous cell carcinoma of sinus, the skin or of the salivary glands
* Stage I cancer
* Radiotherapy planned on primary tumor only, or on neck nodes only. For patients with metastatic lymph nodes from unknown primary head and neck squamous cell carcinoma, patients will be excluded if head and neck mucosa (oropharynx, larynx, hypopharynx) is not included as a target volume for radiotherapy
* Prior radiotherapy of head and neck area
* Concurrent chemotherapy or immunotherapy or hormonotherapy
* Induction chemotherapy
* Concomitant infection requiring IV antibiotics
* cancer other than head and neck cancer within the previous 5 years (baso cellular skin carcinoma and cervix carcinoma excepted)
* conditions that could lead to bad compliance

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Locoregional control | 6 months
  Patient alive with locoregional control at 6 months after the end of radiotherapy

SECONDARY OUTCOMES:
Acute toxicity | 3 months
  Acute toxicity according to the CTC NCI V4 - rate of toxicity by type and by grade
Late toxicity | 18 months
  Late toxicity according to the RTOG late toxicity scale - rate of toxicity by type and by grade
Autonomy | 18 months
  Autonomy according to ADL scale
Health related quality of life | 18 months
  Quality of life according to EORTC QLQ-C30 and QLQ-HN35
Overall survival | 18 months
  Overall survival
Locoregional progression | 18 months
  Locoregional progression
metastasis progression | 18 months
  metastasis progression
Progression free survival | 18 months
  Progression free survival

CONTACTS AND LOCATIONS:
Locations (2):
- Institut Gustave Roussy, Villejuif, France
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: Yes
Data Monitoring Committee will meet every year either by a physical meeting or by conference call. Data on the recruitment, toxicity and autonomy are submitted every year.

REFERENCES:
- See also: GORTEC — http://www.gortec.fr/